CLINICAL TRIAL: NCT03111576
Title: Assessment ofMaternal and FetalVascular Changes inNormotensive andPre-Eclamptic Patients and Its Impact on Pregnancy Outcome.
Brief Title: Vascular Changes in Pre-Eclamptic Patients and Its Impact on Pregnancy Outcome.
Acronym: PE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Assistant professor of Obstetrics and Gynecology, Beni-Suef University
Other Study IDs: Beni-Suef 11
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normotensive: This group will include 50 pregnant women with normal blood pressure between 28 and 34 weeks.
- Pre-eclamptic: This group will include 50 pregnant women with diagnosis of pre-eclampsia between 28 and 34 weeks.

SUMMARY:
Normal pregnancy is associated with vasodilation and decreased peripheral resistance, which is detected as early as 5 weeks' gestation .

Pre-eclampsia is a multi-system disorder of the second half of pregnancy , which is characterized by increased vascular reactivity and peripheral resistance with pathological changes that are consistent with impaired blood flow to the affected vascular beds. Investigators will evaluate fetal and maternal vascular changes in normotensive and pre-eclamptic patients by Ultrasound and Doppler and their impact on prediction of pregnancy outcome.

DETAILED DESCRIPTION:
Pre-eclampsia affects 2-8% of all pregnancies, although treatment is generally effective. However, 10-15% of direct maternal deaths are associated with Pre-eclampsia and eclampsia(WHO, 2011). There is a considerable evidence that generalized endothelial dysfunction underlies the clinical manifestations of the disease (Oladipupo et al., 2014).

It has been demonstrated that peripheral nutritive blood flow is impaired in pregnancies complicated by pre-eclampsia and precedes onset of the disorder (Kenny et al., 2014).

The pathophysiological mechanism is characterized by a failure of the trophoblastic invasion of the spiral arteries which may be associated with an increased vascular resistance of the uterine artery and a decreased perfusion of placenta. (Al-Jameil et al ; 2014 ) Ultrasound of the brachial artery, and Doppler ultrasound of the carotid artery and uterine artery are propaedeutic , non-invasive methods that contribute to the understanding of the pathophysiology of PE and Eclampsia (Takata et al., 2002 ).

Doppler assessment of the placental circulation plays an important role in screening for impaired placentation and its complications of preeclampsia, intrauterine growth restriction and perinatal death. Assessment of the fetal circulation is essential in the better understanding of the pathophysiology of a wide range of pathological pregnancies and their clinical management(Ghidini & Vergani, 2012).

ELIGIBILITY:
Inclusion Criteria:

1. All women will be :

   * Nonsmokers,
   * Nondiabetic,
   * With no family history of vascular diseases.
2. Gestational age at enrolment >28 and <34 weeks of gestation.
3. Singleton pregnancy.
4. Informed consent.
5. 50 Normotensive pregnant women without complications will be defined as controls.
6. 50 Pre-eclamptic patients.

Exclusion Criteria:

* 1. Patients who presented to labor and delivery were excluded as subjects. 2. Growth-restricted fetus due to:

  * marginal insertion of the umbilical cord,
  * placental infarction,
  * fetal minor heart anomaly,
  * Fetal viral infection. 3. Refusal of patient to participate in the study. 4. Multiple gestations. 5. Autoimmune diseases 6. Previous history of PE or IUGR.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: on 50 normotensive pregnant women and 50 Pre-eclamptic patients will attend the antenatal clinic in the obstetric ward in the department of Obstetrics and Gynecology in Benisuef general hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Vascular changes by Doppler imaging | >28-<34 weeks
  Doppler imaging will be undertaken for assessing fetal umbilical, middle cerebral arteries in addition to ductus venosus. Concerning maternal vessel assessment, Doppler will be done for uterine arteries, common carotid and brachial arteries.

SECONDARY OUTCOMES:
Pregnancy outcome | Date of delivery and within 40 days after delivery
  Maternal delivery mode and any complications together with fetal growth restriction or neonatal complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Nesreen Abdel Fattah Abdullah Shehata, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No